CLINICAL TRIAL: NCT05999500
Title: Temple Stay Improves Intestinal Microbiome Profile in Patients With Irritable Bowel Syndrome
Brief Title: The Effectiveness of Temple Stay in Irritable Bowel Syndrome
Status: Recruiting | Type: Observational
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Sang Hoon Kim, Assistant professor, Chung-Ang University
Other Study IDs: TEMPLE
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Irritable Bowel Syndrome; Microbial Colonization
MeSH Terms: conditions — Irritable Bowel Syndrome; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Irritable bowel syndrome patients participating in temple stay: We plan to observe a group of patients aged 20-69 with diarrhea-predominant irritable bowel syndrome who have voluntarily agreed to participate in a temple stay for up to 8 days. Observations will be made before the temple stay, immediately after, and then followed up for 4 weeks after the experience.
  Interventions: Behavioral: Temple stay experience

INTERVENTIONS:
Behavioral: Temple stay experience — Temple stay experience includes diet and behavior changes, such as vegetarian meals (ex. Balwoo Gongyang), mindful eating, no overeating, meditation, participation in daily monastic tasks.

SUMMARY:
This research is a clinical trial aimed at improving the gut microbiome of patients with Irritable Bowel Syndrome (IBS) through a temple stay experience.

Participants in the study are expected to participate in a temple stay experience for a maximum of 8 days. During the temple stay experience, participants are required to fill out a daily symptom questionnaire related to irritable bowel syndrome and record their diet and bowel movements using a dedicated mobile application. Upon completion of the temple stay, participants will conduct an evaluation of personal satisfaction with the experience.

Through this, the study aims to collect and analyze data related to the Templestay experience with the goal of improving the gut microbiome of patients with IBS.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a syndrome characterized by recurrent abdominal pain accompanied by abdominal discomfort, changes in bowel habits, and abdominal bloating. It is a common condition, affecting approximately 10% of the population in Korea, and its chronic gastrointestinal symptoms significantly impact patients' daily life and quality of life.

Factors such as changes in the intestinal microbiota and the intestinal ecosystem are crucial in its etiology. Modern individuals, who are often exposed to numerous stressors, frequently experience persistent intestinal hypersensitivity and inflammation. Foods that are not well digested and fermented in the intestines, producing a significant amount of gas - such as those rich in seasonings, dairy products, caffeine, and alcohol - are known to trigger symptoms. Therefore, it is suggested that a controlled environment like a Temple Stay, which provides both dietary regulation and stress control, could lead to meaningful symptom improvement. However, there is currently a lack of objective scientific research on this.

Our research team hypothesizes that a Temple Stay experience of more than a week could consistently change the microbiome and stabilize psychosocial factors. This might control chronic intestinal inflammation and hypersensitivity, leading to subjective symptom improvement and enhanced treatment satisfaction for patients.

Through this study, we aim to validate the hypothesis that the dietary changes in a Temple Stay environment will drastically alter patients' dietary intake, enrich the composition of the gut microbiome, and consequently reduce the symptoms of IBS, thereby improving the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-69 with diarrhea-predominant irritable bowel syndrome

Exclusion Criteria:

* Monk
* history of irritable bowel syndrome (constipation-predominant), history of inflammatory bowel disease, history of colorectal cancer, history of gastrointestinal resection,
* abnormal blood test (liver function test: AST or ALT more than 1.5 times the normal limit, total bilirubin increase of more than 1.5mg/dL, CCr < 30 mL/min, platelets less than 100,000, PT/aPTT increase of more than 20% of the normal upper limit),
* uncontrolled hypertension and diabetes

Ages: 20 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 20-69 with diarrhea-predominant or constipation-predominant irritable bowel syndrome.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
IBS-SSS | before the event, during the event, 4-weeks after the event
  symptom score for irritable bowel syndrome

SECONDARY OUTCOMES:
Fecal microbiome | before the event, during the event, 4-weeks after the event
  Fecal microbiota composition, microbiome, diversity, Difference in the proportion of the species of primary interest

CONTACTS AND LOCATIONS:
Overall Officials: Jun Kyu Lee, Prof., Principal Investigator — DongGuk University
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Conditionally considering upon reasonable request.